CLINICAL TRIAL: NCT02244762
Title: Evaluation of the Effect of Renal Impairment on the Pharmacokinetics and Metabolism of Hydrocodone and Its Metabolites Following Administration of Hydrocodone Bitartrate Extended-Release (HC-ER) 20 mg Capsules
Brief Title: Pharmacokinetics and Metabolism of Hydrocodone Bitartrate Extended-Release (HC-ER) in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZX002-1002
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2014-09

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild Renal Impairment (Experimental): 20 mg HC-ER
  Interventions: Drug: 20 mg HC-ER
- Moderate Renal Impairment (Experimental): 20 mg HC-ER
  Interventions: Drug: 20 mg HC-ER
- Severe Renal Impairment (Experimental): 20 mg HC-ER
  Interventions: Drug: 20 mg HC-ER

INTERVENTIONS:
Drug: 20 mg HC-ER — 1-72 hours
  Other Names: Zohydro ER
  Arms: Mild Renal Impairment
Drug: 20 mg HC-ER — 1-72 hours
  Other Names: Zohydro ER
  Arms: Moderate Renal Impairment
Drug: 20 mg HC-ER — 1-72 hours
  Other Names: Zohydro ER
  Arms: Severe Renal Impairment

SUMMARY:
Determine the influence of renal impairment on the pharmacokinetics and metabolism of Hydrocodone Bitartrate Extended-Release (HC-ER) 20 mg capsules

DETAILED DESCRIPTION:
Pharmacokinetics and relative bioavailability of hydrocodone and its metabolites under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

All renal-impaired subjects must have meet all of the following inclusion criteria to be eligible to be enrolled into this study. Subjects were eligible for the study if they meet all of the following criteria:

1. Male or non-pregnant, non-lactating females.
2. Subjects were 18-80 years old.
3. Subjects must have had a clinical diagnosis of chronic renal impairment for duration of at least 6 months classified as mild, moderate or severe per Cockcroft Gault criteria (see Appendix A)
4. Renal insufficiency should have been stable with no acute episodes of illness within the previous 2 months due to deterioration of renal function due to any etiology.
5. Female subjects of childbearing potential including those who had a tubal ligation surgery but excluding those who have not experienced a menstrual period for a minimum of 2 years, must have had a negative pregnancy test at the Screening and Day -1 visits, and must consent to use a medically-acceptable method of contraception throughout the entire study period and for 1 week after the study is completed. Medically acceptable methods of contraception include but were not limited to abstinence, birth control pills or patches, vaginal rings, diaphragm with vaginal spermicide, intrauterine device (IUD), and progestin implant or injection (used consistently for 3 months prior to study dosing).
6. Subjects must have voluntarily provided written informed consent.
7. Subjects, in the Investigator's opinion, must have been able to complete all study procedures.

All healthy control subjects must have meet all renal subject inclusion criteria as outlined above with the exception of Inclusion Criteria 2 and 3 which should be substituted with the following to be enrolled into the study:

2a. Must have matched by age (± 10 years) and BMI (±10% of BMI) with some consideration for race and gender to subjects with renal impairment.

3b. Were medically healthy with no clinically significant abnormalities in their laboratory profile as deemed by the investigator.

Exclusion Criteria:

Subjects were not be eligible for the study if they meet any of the following criteria:

1. Women who were pregnant or breastfeeding.
2. Any clinically significant condition that would, in the opinion of the Investigator, preclude study participation.
3. Uncontrolled blood pressure, i.e., subjects has a sitting systolic blood pressure >180 mmHg or <90 mmHg, and/or a sitting diastolic blood pressure >120 mmHg or <50 mmHg at screening.
4. A Body mass Index (BMI) >40 kg/m2.
5. A known allergy or hypersensitivity to hydrocodone, or other opioids.
6. Have taken any investigational drug within 30 days prior to the Day 1 visit or be currently enrolled in another investigational drug study.
7. Have used a monoamine oxidase inhibitor within 14 days prior to the Day 1 visit.
8. Were taking opioids during the 30 days prior to Day 1 or needing to take opioids during the study period.
9. Positive for HIV. Healthy control subjects must have not been Hepatitis C Virus (HCV) positive, renal-impaired subjects can be HCV positive but should not be receiving treatment.
10. A history of any illicit substance abuse in the past 2 years or any history of opioids abuse. Subjects should not have been current abusers of alcohol and must have a negative serum alcohol at Screening and Day-1.
11. Had a positive quantitative urine drug screen for illicit drugs, or non-prescribed controlled substances at screening.
12. Had made a plasma donation within 7 days prior to Day 1.
13. Had made any significant donation or loss of blood within 56 days prior to Day 1.
14. Had taken CYP2D6 and/or 3A4 inhibitors within 7 days prior to Day 1 and/or CYP2D6 and/or 3A4 inducers within 21 days prior to Day 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of hydrocodone and its metabolites of 20 mg HC-ER | Day 1-3
  PK parameters including Cmax, Tmax, , AUC 0-t, AUC 0-inf, T1/2 and Kel

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lasseter, MD, Study Director — Zogenix, Inc.